CLINICAL TRIAL: NCT00795522
Title: An Open-Label Study of the Effects of Desloratadine (Aerius.) Treatment on the Quality of Life of Patients With Chronic Idiopathic Urticaria
Brief Title: An Open-Label Study of the Effects of Desloratadine (Aerius.) Treatment on the Quality of Life of Patients With Chronic Idiopathic Urticaria (Study P02540)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02540
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Desloratadine
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — Subjects will receive DL 5 mg daily for 28 days. Each active DL tablet contains 5 mg of desloratadine
  Other Names: SCH 034117

SUMMARY:
This open-label study is being conducted to determine the effect of DL treatment for CIU on symptom and disease severity, quality of life, daytime functioning, and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >= 18 years of age, of either sex and any race.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation). Women of childbearing potential should be counseled in the appropriate use of birth control while in this study. Women who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.
* Subjects must be in general good health; i.e., they must be free of any clinically significant disease (other than CIU) that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and agree to complete the questionnaires and to record symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary.
* Subjects must have at least a 6-week history of CIU (pruritus and hives) prior to Visit 1 (Screening).
* Subjects must have a pruritus score >= 2 and a hive score >= 1 at Visit 1.
* Subjects must be experiencing a current CIU flare of at least 3 weeks duration, with hives present at least 3 days per week, prior to Visit 1 (Screening).
* Subjects must score the overall condition of CIU >= 2 at both Visit 1 (Screening) and Visit 2 (Baseline).
* Subjects must have a total pruritus score of >= 14 for the sum of morning and evening (reflective) diary scores for the 3 days prior to Visit 2 (Baseline) plus the morning score on the day of Visit 2.
* Women of childbearing potential must have a negative urine pregnancy test at Visit 2 (Baseline).

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications outlined.
* Subjects with asthma requiring chronic use of inhaled or systemic corticosteroids.
* Subjects with drug or food allergies that manifest as skin reactions.
* Subjects with urticaria that is primarily due to physical urticaria or other known etiology.
* Subjects with CIU unresponsive to antihistamines.
* Subjects who have been hospitalized (including an emergency department visit) because of deterioration in their CIU within 3 months prior to Visit 1 (Screening).
* Subjects with a history of hypersensitivity to desloratadine or any of its excipients.
* Subjects previously randomized into this study.
* Subjects who are staff personnel directly involved with the administration of this study.
* Subjects who have any clinically significant metabolic, cardiovascular, immunologic, neurologic, hematologic, gastrointestinal, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect subject safety.
* Subjects with a history of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study.
* Subjects with a history of noncompliance with medications or treatment protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-07; Primary Completion 2005-02 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Short Form 12 (SF-12) Health Survey Questionnaire, mental, physical and total scores on treatment days 7, 14, 21, and 28. | treatment days 7, 14, 21, and 28

SECONDARY OUTCOMES:
Change from Baseline in work/school attendance and self-assessed productivity as measured by the WPAI questionnaire | treatment days 7, 14, 21, and 28
Change from Baseline in pruritus, the number of hives and the maximum size of hives, sleep quality, and activity impairment | treatment weeks 1, 2, 3, and 4
The percent of subjects who rate their response to therapy as either Complete, Marked, or Moderate Relief | day 28